CLINICAL TRIAL: NCT03734172
Title: Rapid and Accurate Diagnosis of Paediatric (RaPaed) TB - An AIDA (Assessment of Innovative Diagnostics and Algorithms for Early and Sensitive Detection of Acute TB) Platform Study
Brief Title: Rapid and Accurate Diagnosis of Paediatric TB (RaPaed-AIDA-TB)
Acronym: RaPaed
Status: Completed | Type: Observational
Sponsor: Michael Hoelscher (Other)
Collaborators: University of Cape Town Lung Institute (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Kamuzu University of Health Sciences (Other); Karolinska Institutet (Other); Research Center Borstel (Other); University of Stellenbosch (Other); Beckman Coulter, Inc. (Industry); Cepheid (Industry); Otsuka Novel Products GmbH (Industry); University of Melbourne (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); National Institute for Medical Research, Tanzania (Other Government); Christian Medical College, Vellore, India (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof Dr med / Sponsor Responsible Person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-AIDA-02
Record Dates: First submitted 2018-06-22; First posted 2018-11-07 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis; Diagnoses Disease
Keywords: Tuberculosis; Paediatrics; Diagnostics
MeSH Terms: conditions — Tuberculosis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Molecular speciation test; Mycobacterial DNA extraction will be performed centrally on stored samples and will be further analysed using classical molecular MTB typing methods (genotyping) as well as by next generation sequencing (genome sequencing).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric diagnostic group: Paediatric diagnostic group
  Interventions: Diagnostic Test: Sample collection

INTERVENTIONS:
Diagnostic Test: Sample collection — Specimen collection

SUMMARY:
This study will serve as a platform to evaluate new diagnostics in children suspected to have TB, establish diagnostic performance (sensitivity and specificity) and calculate positive and negative predictive values in a real-life cohort.

Finally, this study will comprise the results of several tests in its database. This will allow simulation of diagnostic algorithms, that may be composed of screening (i.e. rule-out) tests together with confirmatory tests to maximize sensitivity and specificity.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major cause of child morbidity and mortality in the world. There are an estimated one million new paediatric cases and at least 239.000 deaths per year. As childhood mortality on TB treatment is low at 1%, this highlights the fact that a large proportion of cases are never diagnosed and thereby never receive appropriate treatment.

The inability to correctly and timely diagnose paediatric TB is the main obstacle to controlling disease and preventing adverse outcomes, specifically among infants and young children, children with malnutrition, HIV infection, and drug-resistant TB. Paediatric samples, which are difficult to obtain, have small volumes and low bacterial burden, leading to the low sensitivity of currently applied diagnostic tests for TB, which are geared towards adults.

The World Health Organization has clearly stated that new and improved diagnostics for children are a top priority.

With RaPaed TB, the Sponsor (LMU) designed a project that is ideally suited to evaluate a range of novel diagnostics and sampling strategies in a population of symptomatic children with presumptive TB with a high likelihood of mycobacteriological confirmation of disease. The key aspects of this project are a multi-site collaboration of five geographically distinctive sites in highly TB endemic settings allowing a large sample size, and a high proportion of bacteriologically confirmed cases and making study findings generalizable.

Internationally recognized experts in child TB clinical research are included in the study; FIND's panel of diagnostic tests and expertise in diagnostics development and evaluation as well in the WHO submission and review process of the gathered data; LMU with its track record of delivering high-quality studies in the TB field; two large industry partners dedicated to the development of robust point-of-care assays; and finally, early involvement of National TB Programmes in the studies which will not only add to local capacity development, but also enable rapid local approval and uptake.

974 paediatric patients were enrolled into the RaPaed study in the four African and one Indian sites, with an average confirmation rate of 24% (study target: 25%).

Ten new diagnostic techniques suitable for children are being assessed in this study. These include a new stool protocol and Nasopharyngeal Aspirate for Xpert® MTB/RIF Ultra, TAM-TB from the University of Munich/Beckman Coulter Inc., a host biomarker panel by the University of Stellenbosch, host RNA tests, host protein biomarker tests (i.e. FIND and SomaLogic's host-response serum markers), and two novel urinary LAM tests (i.e. UriTB direct, FUJIFILM-urinary-LAM), and Cepheid's Fingerprick test.

It is realistic to think that this study will lead to WHO endorsement or recommendation of at least two or more new assays or sampling strategies; with FIND leading the WHO submission process which could therefore impact childhood TB policies globally.

In this third period of the RaPaed-TB study, all relevant study documents have been maintained such as the protocol, the Manual of Procedures, SOPs and Worksheets for collecting the data.

Ethics approval for the study conduct and all updates have been obtained centrally and in all study sites by the time of submission of this report.

The database has been maintained and updated, fulfilling its function for study data collection and analysis, as well as enabling study oversight and quality control.

ELIGIBILITY:
Inclusion Criteria:

1. Consent and Assent (if applicable): signed written consent/assent, or witnessed oral consent/assent in the case of illiteracy, before undertaking any study-specific activity. The age threshold for child assent requirement will be laid down in each the Investigator Site File based on the local Ethics Committee requirement.

   Of the following, either criterion 2), OR criterion 3), or both, have to be met:
2. Confirmation of TB disease: microbiological confirmation of active TB disease by positive smear AND/OR culture AND/OR PCR (e.g. GeneXpert®); e.g. in a non-study health facility AND/OR
3. Signs and Symptoms: suspicion of active TB disease (one or more criteria):

   1. Chest X-ray suggestive of TB: cavity AND/OR hilar/mediastinal lymph node enlarged AND/OR military pattern
   2. Weight loss or failure to thrive within the previous 3 months that, in the investigator's opinion, is not solely due to inadequate feeding; or to another non-TB cause.
   3. Any cough combined with loss of weight
   4. Cough alone: duration of > 14 days
   5. Repeated episodes of fever within 14 days not responding to course of antibiotics AND positive TST or IGRA, (for malaria endemic areas: AND after malaria has been excluded by at least a negative rapid test)*
   6. Signs & symptoms of extrapulmonary TB:

      * Enlarged lymph nodes for > 2 weeks, not painful to palpation;
      * Gibbus (especially of recent onset)
      * Non-painful enlarged joint
      * Pleural effusion
      * Pericardial effusion
   7. CSF examination findings in line with TB meningitis with at least elevated protein and low glucose (in relation to serum glucose); OR signs and symptoms in line with TB meningitis/CNS TB if lumbar puncture is contraindicated, in the view of the investigator:

At least one of the following two:

* palsy of oculomotoric nerves of recent onset
* focal neurological symptoms indicating elevated intracranial pressure OR CNS lesions, of recent onset

AND/OR at least two of the following less specific signs of TB meningitis/CNS TB (for malaria endemic areas: AND a negative malaria rapid diagnostic test*):

* Lethargy
* Convulsion
* Meningism (neck stiffness)
* Headache (*the requirement of negative MRDT may be dropped in agreement with the sponsor during study conduct.)

Exclusion Criteria:

1. Critical condition (if study procedures seems like an undue risk to patient's life), such as hypovolemic shock or clinically relevant anaemia (tachypnoea, tachycardia)
2. Body weight is less than 2 kg
3. Children of 15 years of age or older
4. Are currently receiving anti-TB drug(s): ideally, eligible patients should not have received any anti-TB treatment. In exceptions, up to three daily doses given since treatment start before first study blood draw are acceptable for study inclusion

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 14 years old or younger with a suspicion of active TB are eligible for recruitment into the study, if they meet the specified inclusion criteria, and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 974 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificit of new test candidates; against a clinica/microbiological reference standard case definition | 6 months
  The case definition has been defined by an NIH-convened expert panel, published in 2012 and updated in 2015 (S. Graham et al.; CID). This definition describes the diagnostic certainty for a child to suffer from TB.
  Possible classifications:
  * Confirmed active tuberculosis
  * Unconfirmed tuberculosis
  * Unlikely tuberculosis
  This case definition will be made based on the following:
  * Confirmed active tuberculosis: bacteriological confirmation obtained (TB lab; positive culture AND/OR WHO endorsed PCR).
  * Unconfirmed tuberculosis: bacteriological confirmation NOT obtained AND at least two of the following:
  Symptoms suggestive of TB X-ray suggestive of TB Close exposure to TB Positive response to TB treatment
  • Unlikely tuberculosis: defined as bacteriological confirmation NOT obtained AND criteria for "unconfirmed tuberculosis" NOT met

OTHER OUTCOMES:
Ability of new tests to measure response to TB treatment, by measuring the change in experimental test readout over time while receiving TB treatment | 6 months
  Rate of change of new test readout (e.g. antigen detection rates), in children who receive TB treatment
Proportion of children with confirmed TB, and with other diseases, who have acute and chronic lung impairment using spirometry | 12 months
  Spirometry parameters: forced vital capacity (FVC) in l; forced expiratory volume in 1 second (FEV 1)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Professor, Principal Investigator — University Hospital, LMU Munich; Norbert Heinrich, MD, Study Director — University Hospital, LMU Munich
Locations (5):
- Christian Medical College, Vellore, Tamil Nadu, India
- University of Malawi College of Medicine, Blantyre, Malawi
- Centro de Investigação e Treino em Saúde da Polana Caniço, Maputo, Mozambique
- University of Cape Town Lung Institute (UCTLI), Cape Town, Cape, South Africa
- NIMR - Mbeya Medical Research Programme, Mbeya, Tanzania

REFERENCES:
- [Derived] Olbrich L, Nliwasa M, Sabi I, Ntinginya NE, Khosa C, Banze D, Corbett EL, Semphere R, Verghese VP, Michael JS, Graham SM, Egere U, Schaaf HS, Morrison J, McHugh TD, Song R, Nabeta P, Trollip A, Geldmacher C, Hoelscher M, Zar HJ, Heinrich N; RaPaed-AIDA-TB Consortium. Rapid and Accurate Diagnosis of Pediatric Tuberculosis Disease: A Diagnostic Accuracy Study for Pediatric Tuberculosis. Pediatr Infect Dis J. 2023 May 1;42(5):353-360. doi: 10.1097/INF.0000000000003853. Epub 2023 Feb 16. PMID 36854097